CLINICAL TRIAL: NCT04279561
Title: Effects of Novel Androgen Receptor Signaling Inhibitors on PSMA PET Signal Intensity in Patients With Castrate-Resistant Prostate Cancer: A Prospective Exploratory Study
Brief Title: Effect of Androgen Receptor Signaling Inhibitors on 68Ga-PSMA-11 PET/CT Imaging in Patients With Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-002024; NCI-2020-00239 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (68GA-PSMA-11 PET/CT) (Experimental): Patients receive 68Ga-PSMA-11 IV. After 50-100 minutes, patients undergo PET/CT over 20-50 minutes. Patients undergo 68Ga-PSMA-11 PET/CT at baseline, at 1 week and 3 months after initiation of ARSI, and at time of biochemical progression (within 1 year if applicable).
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68 Gozetotide; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo 68Ga-PSMA-11 PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo 68Ga-PSMA-11 PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies the effect of androgen receptor signaling inhibitors on 68Ga-PSMA-11 PET/CT imaging in patients with castration-resistant prostate cancer that has spread to other places in the body (metastatic). Diagnostic procedures, such as 68Ga-PSMA-11 PET/CT, may help in learning how well androgen receptor signaling inhibitors work in killing castration-resistant prostate cancer cells and allow doctors to plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate short- and long-term prostate specific membrane antigen (PSMA) imaging changes in response to androgen receptor signaling inhibitors (ARSI).

SECONDARY OBJECTIVES:

I. To correlate PSMA imaging changes with prostate specific antigen (PSA) kinetics.

II. To correlate PSMA imaging changes with progression free survival. III. To evaluate the changes in PSMA PET staging (miTNM Prostate Cancer Molecular Imaging Standardized Evaluation [PROMISE] criteria) under ARSI.

OUTLINE:

Patients receive gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) intravenously (IV). After 50-100 minutes, patients undergo positron emission tomography (PET)/computed tomography (CT) over 20-50 minutes. Patients undergo 68Ga-PSMA-11 PET/CT at baseline, at 1 week and 3 months after initiation of ARSI, and at time of biochemical progression (within 1 year if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer
* Know metastatic disease on previous imaging, or PSA value ⩾ 1 ng/ml;
* Castration resistant disease with confirmed testosterone level =< 50 ng/ml under prior first-line androgen deprivation therapy (ADT)
* New planned treatment with enzalutamide or abiraterone, darolutamide or apalutamide
* Willingness to undergo ARSI throughout the duration of the study as prescribed by the treating uro-oncologist
* Stated willingness to comply with continuation of ARSI treatment for the duration of the study
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Inability to provide written informed consent
* Known inability to remain still and lie flat for duration of each imaging procedure (about 30 minutes)
* Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy
* A baseline superscan pattern on bone scan
* Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, patients with a prior history of malignancy that has been adequately treated and who have been disease free for more than 3 years are eligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in 68Ga-PSMA-11 lesion and total-body uptake (standardized uptake value [SUV]max and SUVmean) over time in response to androgen receptor signaling inhibitors (ARSI) | Baseline, assessed up to 1 year
  Changes are expressed in terms of percentage changes from baseline positron emission tomography (PET) (before ARSI). Will utilize mixed effect regression models to evaluate the change over time in PSMA results.

SECONDARY OUTCOMES:
Prostate specific antigen (PSA) kinetics under ARSI | Baseline, assessed up to 1 year
  Comparison of 68Ga-PSMA-11 uptake (SUVmax and SUVmean) changes over time to PSA kinetics under ARSI. Will use mixed effects regression models to correlate the PSMA and PSA time trends. These models will include the effect of time and the PSMA by time interaction effect.
Biochemical progression free survival (bPFS) | Up to 1 year
  Correlation between 68Ga-PSMA-11 uptake (SUVmax and SUVmean) changes and time of bPFS under ARSI. Will utilize Cox-proportional hazards regression models. PSMA results will be treated as a time dependent covariate in these models.
Changes in lesion size on cross sectional imaging under ARSI | Up to 1 year
  Correlation between SUVmax from 68Ga-PSMA-11 PET and lesion size on cross sectional imaging under ARSI.
Changes in staging (PSMA miTNM PROMISE criteria) under ARSI | Up to 1 year
  Will utilize mixed effects regression models to evaluate the change in staging over time.
Incidence of adverse events | Up to 1 year
  Assessed by Common Terminology Criteria for Adverse Events 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Sonni I, Gafita A, Unterrainer LM, Alano RM, Lira S, Shen J, Drakaki A, Grogan T, Rettig MB, Czernin J, Calais J. Effects of novel androgen receptor signaling inhibitors on PSMA PET signal intensity in patients with castrate-resistant prostate cancer: a prospective exploratory serial imaging study. EJNMMI Res. 2023 Oct 30;13(1):95. doi: 10.1186/s13550-023-01048-4. PMID 37902861